CLINICAL TRIAL: NCT02628652
Title: A Randomised, Single-Blind, Controlled Study to Evaluate the Tolerability of Prebiotics on the Microbiota
Brief Title: Study to Evaluate the Tolerability of Prebiotics on the Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AFCRO-057
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Microbiome; FOS; polyglycan; prebiotic; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Gluco-Galacto-Oligosaccharide (GOS) (Experimental): Subjects randomized to this treatment arm will ingest GOS once per day for a total of 14 days. One level of GOS will be taken during Phase I and 2 levels of GOS will be taken during Phase II.
  Interventions: Dietary Supplement: GOS
- Gluco-Oligosaccharide (GLOS) (Experimental): Subjects randomized to this treatment arm will ingest GLOS once per day for a total of 14 days. One level of GLOS will be taken during Phase I and 2 levels of GLOS will be taken during Phase II.
  Interventions: Dietary Supplement: GLOS
- FructoOligosaccharide (FOS) (Active Comparator): Subjects randomized to this treatment arm will ingest FOS once per day for a total of 14 days. One level of FOS will be taken during Phase I and 2 levels of FOS will be taken during Phase II.
  Interventions: Dietary Supplement: FOS

INTERVENTIONS:
Dietary Supplement: GOS
  Arms: Gluco-Galacto-Oligosaccharide (GOS)
Dietary Supplement: GLOS
  Arms: Gluco-Oligosaccharide (GLOS)
Dietary Supplement: FOS
  Arms: FructoOligosaccharide (FOS)

SUMMARY:
The primary objective of this study is to determine the tolerability of two polyglycan food ingredients, GOS and GLOS, at two different levels in healthy human subjects. The comparator in this study will be Inulin FOS, a commercially available glycan supplement.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent,
2. Be male or female, between 18 and 40 years of age,
3. Have a BMI ≥ 20 & ≤ 27 kg/m2,
4. Be a non-pregnant female,
5. Be in generally good health,
6. Subjects will continue on his/her normal diet and exercise routine,
7. Be an Irish National.

Exclusion Criteria:

1. Are less than 18 and greater than 40 years of age,
2. Females are pregnant, lactating or wish to become pregnant during the study. Female subject is currently either of:

   * non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or any female who is surgically sterilized (via documented hysterectomy or bilateral tubal ligation). (For purposes of this study, postmenopausal is defined as one year without menses), OR
   * child bearing potential, the subject is eligible to enter and participate in this study if she is not lactating and has a negative urine pregnancy test at the screening visit, visit 2 and upon completion of the study at visit 7. The subject must also agree to one of the following methods of contraception: i. Complete abstinence from intercourse two weeks prior to administration of study, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study medication in cases where subject discontinues the study prematurely. (Subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit.) or, ii. has a male sexual partner who is surgically sterilized prior to the Screen Visit and is the only male sexual partner for that subject or, iii. sexual partner(s) is of the same gender or, iv. Oral or implant contraceptives (either combined or progestogen only) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm. (Women of child-bearing potential using an oral contraceptive in combination with a double-barrier method of contraception are required to continue to use this form of contraception for 1 week following discontinuation of study medication) or, v. Use of double-barrier contraception, specifically, a spermicide plus a mechanical barrier (e.g. male condom, female diaphragm). The subject must be using this method for at least 1 week following the end of the study or, vi. Use of any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year. The subject must have the device inserted at least 2 weeks prior to the first Screen Visit, throughout the study, and 2 weeks following the end of the study.
3. Are hypersensitive to any of the components of the test product,
4. Are currently taking probiotic or prebiotic supplements, or have taken them in the past 28 days,
5. Unwilling to avoid probiotics/prebiotics supplements for the duration of the study
6. Subject has taken antibiotics in the previous 3 months,
7. Have a significant acute or chronic, unstable and untreated disease or any condition which contraindicates, in the investigators judgement, entry to the study,
8. Subject is a smoker,
9. Subject has a history of drug and/or alcohol abuse at the time of enrolment,
10. Having a condition or have taken a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results;
11. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial,
12. Subjects may not be receiving treatment involving experimental drugs,
13. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study,
14. Have a malignant disease or any concomitant end-stage organ disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events in each group | 28 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials/ University Cork College, Cork, Ireland